CLINICAL TRIAL: NCT06977009
Title: Influence of Occlusal Reduction on Endodontic Postoperative Pain: a Randomized Clinical Trial
Brief Title: Influence of Occlusal Reduction on Endodontic Postoperative Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Abdulrahman Mwaffaq Kahhaleh, Masters studnet, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: occlusal reduction after RCT
Record Dates: First submitted 2025-05-01; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Post Operative Pain Management

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will take place at the postgraduate endodontic clinic department at JU Hospital to assess the effect of occlusal reduction on post-operative pain. Participants will be enrolled from the pool of patients referred to the department of endodontics at JUH for root canal treatment, and the trial will be carried out on those diagnosed with necrotic pulps or previously initiated (accessed) teeth.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- occlusal reduction (Intervention group) (Active Comparator): all occlusal contacts on the functional and non-functional cusps as well as on the marginal ridges will be reduced using a diamond bur.
  Interventions: Procedure: Occlusal Reduction
- no occlusal reduction (Control group) (No Intervention): all occlusal contacts will remain intact.

INTERVENTIONS:
Procedure: Occlusal Reduction — patients will be allocated to either undergo occlusal reduction (Intervention group) where all occlusal contacts on the functional and non-functional cusps as well as on the marginal ridges will be reduced using a diamond bur, or not undergo occlusal reduction (Control group) where all occlusal contacts will remain intact.
  The presence or absence of contact will be confirmed using articulating paper where occlusal surfaces will be dried and articulating paper will be held between the teeth with the mandible guided to the centric position. Intact occlusion will be assessed by examining the marks on the teeth.
  A high-speed handpiece with copious coolant will be used to remove occlusal contacts (Intervention group) or just moved above the surface of the tooth without contacting the occlusal surface (Control group) to facilitate patient blinding.
  Arms: occlusal reduction (Intervention group)

SUMMARY:
This study aims to assess the impact of occlusal reduction on post-operative pain after single-visit root canal treatment in patients with necrotic pulps or previously initiated (accessed).

DETAILED DESCRIPTION:
A randomized clinical trial will take place at the postgraduate endodontic clinic department at JU Hospital to assess the effect of occlusal reduction on post-operative pain. Participants will be enrolled from the pool of patients referred to the department of endodontics at JUH for root canal treatment, and the trial will be carried out on those diagnosed with necrotic pulps or previously initiated (accessed) teeth.

Patients will undergo root canal treatment by postgraduate students, under rubber dam, and using the dental operating microscope.

At the completion of endodontic treatment, the numbered, sealed, randomization envelope will be opened by the operator, and patient allocation will be revealed.

Access cavity will be sealed with Glass ionomer restoration, then patients will be allocated to either undergo occlusal reduction (Intervention group) where all occlusal contacts on the functional and non-functional cusps as well as on the marginal ridges will be reduced using a diamond bur, or not undergo occlusal reduction (Control group) where all occlusal contacts will remain intact.

The presence or absence of contact will be confirmed using articulating paper where occlusal surfaces will be dried and articulating paper will be held between the teeth with the mandible guided to the centric position. Intact occlusion will be assessed by examining the marks on the teeth.

A high-speed handpiece with copious coolant will be used to remove occlusal contacts (Intervention group) or just moved above the surface of the tooth without contacting the occlusal surface (Control group) to facilitate patient blinding.

The patient will be told to not change his or her restoration to a permanent restoration for at least a week (before the completion of data collection).

Treatment will be completed in a single visit.

Pain will be assessed according to a visual analog scale (VAS). Scores will be taken before commencing the procedure (pre-operative pain) and after the treatment at different time intervals; 6, 24, 48 hours, and 1 week after. This will be done by calling the patients by phone to record the degree of pain at these intervals.

The assessment of postoperative pain will be performed by a researcher-examiner blinded to the carried-out treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy subjects (ASA I&II) between the age of 18 and 70 years
2. Patients diagnosed with necrotic pulp or previously initiated (accessed).
3. Posterior maxillary or mandibular molar tooth.
4. Presence of an opposing tooth (or teeth) with normal occlusal contact with the opposing tooth (or teeth).
5. Tooth needs cuspal coverage.

Exclusion Criteria:

1. Pregnant females.
2. Patients with significant medical conditions (ASA III & IV).
3. Reported bruxism or clenching.
4. Took analgesics\antibiotics or other drugs that might alter their pain during the last 12 hours preoperatively.
5. A history of allergic reactions to any of the medications and/or materials used.
6. Patients with a tooth that had no contacts or premature contact, fewer than three teeth on one side of the jaw.
7. Greater than grade I mobility or pocket depth greater than 5mm.
8. Non-restorable crowns, severely curved root canals, or post-treatment endodontic disease were, also, excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
impact of occlusal reduction on post-operative pain after single-visit root canal treatment by using the visual analog scale (VAS). | from the enrollment of the patient up to 1 week for each patient
  to assess the impact of occlusal reduction on post-operative pain after single-visit root canal treatment in patients with necrotic pulps or previously initiated (accessed) by using visual analog scale (VAS) at 6, 24, 48 hours, and 1 week following the treatment.
  The VAS consists of a 10-cm line anchored by two extremes "No pain" and "pain as bad as could be". The patients were asked to choose the mark that represented their level of pain. Pain level was assigned to one of four categorical groups: None (0); Mild (1-3); Moderate (4- 6); Severe (7-10). The scale was explained visually, verbally and numerically to facilitate its use by the participants.
  This will be done by calling the patients by phone to record the degree of pain at these intervals as explained in the study description.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hammad, Associate Professor, Study Director — University of Jordan
Locations (1):
- Jordan university hospital, Amman, Amman Governorate, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shamszadeh S, Shirvani A, Asgary S. Does occlusal reduction reduce post-endodontic pain? A systematic review and meta-analysis. J Oral Rehabil. 2020 Apr;47(4):528-535. doi: 10.1111/joor.12929. Epub 2020 Jan 16. PMID 31880822
- [Background] Nguyen-Nhon D, Nagendrababu V, Pulikkotil SJ, Rossi-Fedele G. Effect of occlusal reduction on postendodontic pain: A systematic review and meta-analysis of randomised clinical trials. Aust Endod J. 2020 Aug;46(2):282-294. doi: 10.1111/aej.12380. Epub 2019 Oct 22. PMID 31638301
- [Background] Parirokh M, Rekabi AR, Ashouri R, Nakhaee N, Abbott PV, Gorjestani H. Effect of occlusal reduction on postoperative pain in teeth with irreversible pulpitis and mild tenderness to percussion. J Endod. 2013 Jan;39(1):1-5. doi: 10.1016/j.joen.2012.08.008. Epub 2012 Sep 29. PMID 23228248
- See also: Effect of Occlusal Adjustment on Postoperative Pain after Root Canal Treatment: A Randomized Clinical Trial — https://doi.org/10.1590/0103-6440202003248